CLINICAL TRIAL: NCT01342016
Title: A Randomized, Double-blind Double Dummy, Parallel Control and Multi-center Clinical Trial to Compare the Efficacy and Safety of Tacrolimus Capsules in Treatment of Lupus Nephritis With Leflunomide Tablets
Brief Title: A Study to Compare the Efficacy and Safety of Tacrolimus Capsules With Leflunomide Tablets in Lupus Nephritis Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to safety concern of active control drug
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F506-CL-0911
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Lupus Nephritis
Keywords: prograf; nephritis; leflunomide; immunosuppressant
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — Tacrolimus; Leflunomide; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tacrolimus group (Experimental): tacrolimus capsule + leflunomide placebo
  Interventions: Drug: tacrolimus capsule; Drug: leflunomide placebo; Drug: prednisone
- leflunomide group (Active Comparator): tacrolimus placebo + leflunomide tablet
  Interventions: Drug: tacrolimus placebo; Drug: leflunomide tablet; Drug: prednisone

INTERVENTIONS:
Drug: tacrolimus capsule — oral
  Other Names: prograf; FK506
  Arms: tacrolimus group
Drug: tacrolimus placebo — oral
  Arms: leflunomide group
Drug: leflunomide tablet — oral
  Other Names: airuohua
  Arms: leflunomide group
Drug: leflunomide placebo — oral
  Arms: tacrolimus group
Drug: prednisone — oral

SUMMARY:
The purpose of this study is to compare the efficacy and safety of tacrolimus capsules with leflunomide tablets in the treatment of lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* body weight 40-100kg
* diagnosed as systemic lupus erythematosus, (according to American College of Rheumatology Diagnostic Criteria,1997)
* diagnosed as type III/ IV of lupus nephritis by renal biopsy within 6 months
* 24hr proteinuria ≥2g and/or active urinary sediments

Exclusion Criteria:

* receiving immunosuppressant
* receiving routine treatment of tacrolimus and leflunomide within 1 month
* receiving nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 months before the study
* history of allergy to tacrolimus and leflunomide
* anticipated maintenance dialysis persisted over 8 weeks; or already being dialyzed over 2 weeks before recruitment
* planning to receive kidney transplantation or in the near future or having a history of undergoing kidney transplantation
* serum creatinine (Scr) ≥3mg/dl or estimated glomerular filtration rate (eGFR) < 30ml/min
* diabetes mellitus patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
remission rate (partial remission + complete remission) | at 6 months after treatment

SECONDARY OUTCOMES:
urinary protein excretion for 24 hrs (24hr proteinuria) | at 12 weeks and 24 weeks
serum albumin level | at 12 weeks and 24 weeks
serum creatinine level | at 12 weeks and 24 weeks
estimated glomerular filtration rate (eGFR) | at 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (12):
- China (12):
  - Beijing
  - Fujian
  - Hubei
  - Hunan
  - Jiangsu
  - Jilin
  - Liaoning
  - Shandong
  - Shanghai
  - Shanxi
  - Sichuan
  - Zhejiang